CLINICAL TRIAL: NCT01191918
Title: A Double-Blind, Placebo-Controlled Evaluation of The Efficacy and Safety of AChE Inhibitor Donepezil As Adjunctive Treatment to Mood Stabilizers in Acute Mania
Brief Title: The Efficacy and Safety of AChE Inhibitor Donepezil As Adjunctive Treatment to Mood Stabilizers in Acute Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: The Davis Foundations (Other)
Responsible Party: Zheng Lu, Shanghai Mental Health Center, Shanghai Jiaotong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zlu001
Record Dates: First submitted 2010-08-29; First posted 2010-08-31 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Bipolar Disorder; Mania
Keywords: acetylcholinesterase inhibitor; donepezil; bipolar disorder; mania; lithium
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Donepezil; Lithium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- donepezil (Experimental): donepezil plus Lithium
  Interventions: Drug: Donepezil and Lithium
- Control (Placebo Comparator): Placebo plus Lithium
  Interventions: Drug: Placebo plus Lithium

INTERVENTIONS:
Drug: Donepezil and Lithium — Donepezil dose will be started at 5mg/d and increased to 10 mg/d in 1 week.
  Other Names: Aricept
  Arms: donepezil
Drug: Placebo plus Lithium
  Arms: Control

SUMMARY:
There is a high rate of partial response to standard thymoleptic medication. In this study the investigators want to evaluate the safety and efficacy of donepezil as adjunctive treatment to mood stabilizers in bipolar disorder with acute mania. The investigators hypotheses were that there would be greater mean reduction in manic symptoms with donepezil augmentation of lithium compared with placebo.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic mental illness that affects 1-2% of the general population. Lithium and valproate are effective for treatment of acute mania for many patients. However up to half of patients do not respond adequately to currently approved treatments in the acute phase of mania. More effective treatment for mania are need. Imbalance in cholinergic and adrenergic tone has long been postulated in the pathophysiology of bipolar disorder. In the pathophysiology of mania,relative cholinergic hypoactivity was being implicated. Donepezil is a centrally acting reversible acetylcholinesterase inhibitor. It is approved for the treatment of Alzheimer's disease. In an open case series with standardized ratings, addition of donepezil 5-10 mg/day to ongoing mood-stabilizer treatment was associated with marked improvement in treatment-resistant mania. We want to conduct a 4-week randomized, double-blind, placebo-controlled trial of donepezil as augmentation of lithium in patients with acute manic episode to evaluate the safety and efficacy of donepezil as adjunctive treatment to mood stabilizers in bipolar disorder with acute mania.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have DSM-IV diagnosis of bipolar disorder with acute manic episode who are admitted as inpatient
2. Young Mania Rating Scale (YMRS) total score >20 (based on mean scores of two ratings after admission)
3. Physical examination, laboratory results (eg.EKG) from screening visit normal, or abnormal clinically insignificant

Exclusion Criteria:

1. Having history of allergy to donepezil or Lithium.
2. Having active suicide or homicide attempt or intent
3. Having severe medical conditions or taking multiple medications for medical conditions
4. Investigational drug treatment within past 30 days
5. Having a drug screen positive for any drug of abuse at screening
6. Self-report of active substance abuse in the past 2 weeks or substance dependence in the past 2 months
7. Diagnosis of schizophrenia, dementia, delirium, seizure disorder, obsessive compulsive disorder, or unstable medical condition
8. Administration of any investigational drug within 30 days of screening
9. Pregnancy or lactation
10. Asthma requiring chronic medication treatment or ongoing use of anticholinergic medications or cholinomimetics
11. Other factors that investigator consider not suitable for the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Total score change of Young Mania Rating Scale | from baseline to week 4
  Patients were assessed by outcomes assessores at 0 hour(h), 2h,4h,6h,8h,10h,12h,24h,1 week (w), 2w, 4w

SECONDARY OUTCOMES:
Treatment Emergent Symptom Scale | from baseline to week4
  assessed at day 1, week1, week 2, week4
Clinical Global Impression | frome baseline to week 4
  assessed at 0h, 2h,4h,6h,8h,10h,12h,24h,week1, week2, week4
Brief Psychiatric Rating Scale | frome baseline to week 4
  assessed at 0h, 2h,4h,6h,8h,10h,12h,24h,week1, week2, week4

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Lu, MD, Principal Investigator — Shanghai Mental Health Center